CLINICAL TRIAL: NCT03011060
Title: A Prospective Randomized Controlled Trail to Evaluate Efficacy and Safety of Sequential Neo-adjuvant Chemotherapy Plus Surgery Followed by Capecitabine Versus Conventional Postoperative Adjuvant Chemotherapy
Brief Title: Sequential Neo-adjuvant Chemotherapy Followed by Capecitabine Vs. Conventional Adjuvant Chemotherapy in Breast Cancer
Acronym: NACVCAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: First Hospital of China Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Qingdao University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Baotou Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLUDBSCRH 001
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Breast Neoplasm Female
Keywords: neo-adjuvant chemotherapy; pathological complete response; Neoadjuvant Therapy; Capecitabine; Chemotherapy, Adjuvant
MeSH Terms: interventions — Induction Chemotherapy; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NAC not achieving pCR (Experimental): Patients in the study group will accept neo-adjuvant chemotherapy. Among these patients, those who do not achieve pCR after neo-adjuvant chemotherapy will be treated with Capecitabine after surgery. And then they will be followed up for 5 years.
  Capecitabine 1000mg/m2 tablets twice a day for 8 cycles.
  Interventions: Procedure: Neo-adjuvant Chemotherapy; Drug: Capecitabine
- NAC achieving pCR (Experimental): Patients in the study group will accept neo-adjuvant chemotherapy. In these patients, those who reach to pCR after neo-adjuvant chemotherapy will be followed up for 5 years after surgery.
  Interventions: Procedure: Neo-adjuvant Chemotherapy
- Adjuvant Chemotherapy (No Intervention): Patients in the control group will accept surgeries and corresponding adjuvant chemotherapy.They will be followed up for 5 years after adjuvant chemotherapy.

INTERVENTIONS:
Procedure: Neo-adjuvant Chemotherapy — A preoperative chemotherapy based on anthracyclines and taxanes.
  Other Names: Preoperative Chemotherapy; Primary Chemotherapy; Induction Chemotherapy
  Arms: NAC achieving pCR; NAC not achieving pCR
Drug: Capecitabine — Capecitabine 1000mg/m2 tablets twice a day for 8 cycles.
  Other Names: Xeloda
  Arms: NAC not achieving pCR

SUMMARY:
This study evaluates whether sequential neo-adjuvant chemotherapy plus surgery followed by Capecitabine could achieve additional benefits over traditional postoperative chemotherapy. In the study group, patients that do not achieve pathological complete response(pCR) will receive sequential neo-adjuvant chemotherapy followed by Capecitabine. In the control group, patients will be treated with postoperative adjuvant chemotherapy.

DETAILED DESCRIPTION:
Neo-adjuvant chemotherapy(NAC) is a standard treatment for locally advanced breast cancer(LABC). By down-staging LABC, NAC is able to make inoperable cases operable as well as to make breast conserving surgery an option again for some patients.Neo-adjuvant chemotherapy is more and more widely used in operable breast cancer since it provides critical information on chemotherapy response. However, only 15% to 20% of the patients can benefit from Neo-adjuvant chemotherapy and achieve pCR. Although we obtained the information chemotherapy response for the rest of the patients who received Neo-adjuvant chemotherapy, there are still controversies on how the information will be used for further treatment. Therefore, it is a problem that needs resolving how these patients can benefit from the information Neo-adjuvant chemotherapy provides and whether Neo-adjuvant chemotherapy can replace conventional adjuvant chemotherapy at all. Our study aims to make Neo-adjuvant chemotherapy benefit more patients.

Registered patients in stage Ⅰ- Ⅲ A breast cancer is randomly split into two groups(study group and control group).In the study group, patients achieving pCR will be followed up for 5 years while patients that do not achieve pCR after neo-adjuvant chemotherapy will be treated with Capecitabine for 8 cycles after surgery. On the other hand, patients in the control group will accept surgeries and conventional adjuvant chemotherapies. Follow-up study will last 5 years. DFS and OS will be compared between the two groups.

This study provides an important basis and methods for the further treatment of patients after neo-adjuvant chemotherapy. It discusses whether neo-adjuvant chemotherapy could replace conventional adjuvant chemotherapy and become a new standard for breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed unilateral invasive carcinoma (all pathological types);
2. No gross or microscopic residual tumor after resection;
3. Clinical stage Ⅰ-stage Ⅲ A, no absolute surgical contraindications;
4. Eastern Cooperative Oncology Group(ECOG) score ≤1;
5. Accepting adjuvant chemotherapy within 15 days after surgery;
6. No peripheral neuropathy;
7. Normal bone marrow and organ functions:

   1. Bone marrow function: ANC≥1500/mm3，PLT≥100000/mm3，HGB≥8g/dl
   2. Renal function: serum creatinine≤1.5 times the upper limit of normal(ULN), Liver function: total bilirubin ≤1.5 times the upper limit of normal，AST≤2.5 times the upper limit of normal，alanine aminotransferase(ALT)≤2.5 times the upper limit of normal
   3. Cardiac function:LVEF≥50%
8. Signed informed consent form.

Exclusion Criteria:

1. Patients with the history of oral fluorouracil chemotherapy or Chinese medicine treatment;
2. Patients with organ dysfunction:

   1. Renal function: serum creatinine>1.5 times the upper limit of normal
   2. Liver function: total bilirubin>1.5 times the upper limit of normal，AST>1.5 times the upper limit of normal, alanine aminotransferase(ALT)>1.5 times the upper limit of normal or alkaline phosphatase (ALP) >2.5 times the upper limit of normal
   3. Cardiac function：LVEF<50%;
3. Human epidermal growth factor receptor-2(HER-2) positive patients who cannot receive Herceptin treatment with a left ventricular ejection fraction(LVEF) less than 55%;
4. Patients allergic to docetaxel, capecitabine, epirubicin and cyclophosphamide;
5. Patients with severe systemic disease and/or uncontrollable infections;
6. Patients with previous malignancies, including contralateral breast cancer;
7. Patients with severe cardiovascular and cerebrovascular disease(i.e. Unstable angina, chronic cardiac failure, uncontrollable high blood pressure of >150/90 mmhg, myocardial infarction and cerebrovascular accident) history within 6 months before randomization;
8. Pregnant or lactating women.
9. Patients who have cognitive or psychological impairment as well as cannot understand the test program or stand side effects, which will result in a suspension of the trial program and follow-up;
10. Patients without personal freedom or independent civil capacity.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1588 (Estimated)
Dates: Start 2016-12; Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | 5 years

SECONDARY OUTCOMES:
Overall survival(OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fan Zhimin, Professor, Study Chair — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fisher B, Brown A, Mamounas E, Wieand S, Robidoux A, Margolese RG, Cruz AB Jr, Fisher ER, Wickerham DL, Wolmark N, DeCillis A, Hoehn JL, Lees AW, Dimitrov NV. Effect of preoperative chemotherapy on local-regional disease in women with operable breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-18. J Clin Oncol. 1997 Jul;15(7):2483-93. doi: 10.1200/JCO.1997.15.7.2483. PMID 9215816
- [Result] Bear HD, Anderson S, Smith RE, Geyer CE Jr, Mamounas EP, Fisher B, Brown AM, Robidoux A, Margolese R, Kahlenberg MS, Paik S, Soran A, Wickerham DL, Wolmark N. Sequential preoperative or postoperative docetaxel added to preoperative doxorubicin plus cyclophosphamide for operable breast cancer:National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2006 May 1;24(13):2019-27. doi: 10.1200/JCO.2005.04.1665. Epub 2006 Apr 10. PMID 16606972
- [Result] Specht J, Gralow JR. Neoadjuvant chemotherapy for locally advanced breast cancer. Semin Radiat Oncol. 2009 Oct;19(4):222-8. doi: 10.1016/j.semradonc.2009.05.001. PMID 19732686
- [Result] Mathew J, Asgeirsson KS, Cheung KL, Chan S, Dahda A, Robertson JF. Neoadjuvant chemotherapy for locally advanced breast cancer: a review of the literature and future directions. Eur J Surg Oncol. 2009 Feb;35(2):113-22. doi: 10.1016/j.ejso.2008.03.015. Epub 2008 May 23. PMID 18502088
- [Result] Mieog JS, van de Velde CJ. Neoadjuvant chemotherapy for early breast cancer. Expert Opin Pharmacother. 2009 Jun;10(9):1423-34. doi: 10.1517/14656560903002105. PMID 19505212
- [Result] Alliot C. In vivo chemosensitivity-adapted preoperative chemotherapy in patients with early-stage breast cancer. Ann Oncol. 2005 Sep;16(9):1559-60; author reply 1560-1. doi: 10.1093/annonc/mdi287. Epub 2005 Aug 3. No abstract available. PMID 16079161
- [Result] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola-Vuorinen A, Tanner M, Asola R, Kokko R, Ahlgren J, Auvinen P, Hemminki A, Paija O, Helle L, Nuortio L, Villman K, Nilsson G, Lahtela SL, Lehtio K, Pajunen M, Poikonen P, Nyandoto P, Kataja V, Bono P, Leinonen M, Lindman H; FinXX Study Investigators. Adjuvant capecitabine in combination with docetaxel and cyclophosphamide plus epirubicin for breast cancer: an open-label, randomised controlled trial. Lancet Oncol. 2009 Dec;10(12):1145-51. doi: 10.1016/S1470-2045(09)70307-9. Epub 2009 Nov 10. PMID 19906561
- [Result] M Toi, S-J Lee.Abstract S1-07: A phase III trial of adjuvant capecitabine in breast cancer patients with HER2-negative pathologic residual invasive disease after neoadjuvant chemotherapy (CREATE-X, JBCRG-04). American Association for Cancer Research 76(4 Supplement):S1-07,2016